CLINICAL TRIAL: NCT01477502
Title: Clinical Value of Homeopathic Assessment and Treatment for Prophylaxis of Recurrent Urinary Tract Infections in Persons With Spinal Cord Injury
Brief Title: Clinical Value of Homeopathic Prophylaxis of Recurrent Urinary Tract Infections in Persons With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011-24; 11050 (Other: Ethical committe of the Kanton Lucerne, Switzerland)
Record Dates: First submitted 2011-11-17; First posted 2011-11-22 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Symptomatic Urinary Tract Infection; Spinal Cord Injury
Keywords: urinary tract infection; spinal cord injury; homeopathy; prevention
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Tract Infections | interventions — Homeopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- individual homeopathic treatment (Active Comparator): participants receive homeopathic treatment in addition to standard prevention measures for UTI
  Interventions: Other: individual homeopathic treatment
- standard prophylaxis (Other)
  Interventions: Other: standard treatment without homeopathy

INTERVENTIONS:
Other: individual homeopathic treatment — participants are diagnosed by a trained homeopath and receive individualized homeopathic treatment in addition to standard UTI prophylaxis
  Arms: individual homeopathic treatment
Other: standard treatment without homeopathy — participants receive standard UTI prophylaxis
  Arms: standard prophylaxis

SUMMARY:
recurrent symptomatic urinary tracts infections (UTI) in persons with spinal cord injury are a frequent problem, leading to significant morbidity and to a decreased quality of life.

* until today, there is no effective prophylaxis for UTI for patients with spinal cord injury.
* homeopathy has been shown to be an effective treatment option in several chronic diseases
* study hypothesis: the addition of homeopathic assessment and treatment to a standard prevention strategy for recurrent UTI will significantly reduce the number of symptomatic UTI per year in this group of patients compared to standard prevention alone

ELIGIBILITY:
Inclusion Criteria:

* neurogenic bladder dysfunction treated by intermittent catheterization
* recurrent (>3/year) symptomatic urinary tract infections

Exclusion Criteria:

* inability to speak German
* already under homeopathic treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
number of symptomatic urinary tract infections | one year

SECONDARY OUTCOMES:
number of symptomatic urinary tract infections compared to the previous year | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Pannek, MD, Principal Investigator — Swiss Paraplegic Center
Locations (1):
- Swiss Paraplegic center, Nottwil, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Pannek J, Pannek-Rademacher S, Jus MS, Wollner J, Krebs J. Usefulness of classical homeopathy for the prophylaxis of recurrent urinary tract infections in individuals with chronic neurogenic lower urinary tract dysfunction. J Spinal Cord Med. 2019 Jul;42(4):453-459. doi: 10.1080/10790268.2018.1440692. Epub 2018 Feb 27. PMID 29485355